CLINICAL TRIAL: NCT01930864
Title: Phase II Trial of Metformin Combined to Irinotecan for Refractory Metastatic or Recurrent Colorectal Cancer
Brief Title: Metformin Plus Irinotecan for Refractory Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: University of Campinas, Brazil (Other); AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MetIri
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms; Adenocarcinoma
Keywords: metformin; colorectal cancer; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma | interventions — Metformin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metfomin + irinotecan (Experimental): Irinotecan 350mg/m² q21d + metformin up to 2500mg/d until disease progression, prohibitive toxicity or consent withdrawal
  Interventions: Drug: metformin; Drug: irinotecan

INTERVENTIONS:
Drug: metformin — metformin up to 2500mg/d
Drug: irinotecan — Irinotecan 350 mg/m² IV q21d

SUMMARY:
MetIri seeks to identify if metformin combined to irinotecan can improve tumor control.

DETAILED DESCRIPTION:
MetIri is a two-stage single arm Phase II assessing the role of combination of metformin to irinotecan for colorectal cancer patients already treat with oxaliplatin, fluoropyrimidine, irinotecan and an anti-EGFr antibody if KRAS wild-type.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Biopsy-proven colorectal adenocarcinoma
* Ineligibility for curative intent therapy, e.g., surgery or radiation
* Disease progression after oxaliplatin (either adjuvant or palliative), fluoropyrimidine (either adjuvant or palliative), irinotecan, and if Kras wild type a anti-EGFR therapy
* Assessable disease according to RECIST v1.1

Exclusion Criteria:

* known hypersensitivity to metformin or irinotecan
* Uncontrolled Central nervous system metastasis
* Acute or chronic severe infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Non-Progression at week 12th of treatment | 12th week
  Non-Progression at week 12th of treatment

SECONDARY OUTCOMES:
Progression-free survival | 12th week
  Progression-free survival
Overall Survival | 12th week
  Overall Survival
Quality of life | 12th week
  Measured by EORTC QLQ C30
Safety | 12th week
  Assessment of toxicity according to CTC 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Joao Paulo SN Lima, MD, PhD, Principal Investigator — AC Camargo Cancer Center
Locations (2):
- Brazil (2):
  - Barretos Cancer Hospital, Barretos, São Paulo
  - State University of Campinas, Campinas, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Upon data collection, the info will be put on a online database

REFERENCES:
- [Background] Rocha GZ, Dias MM, Ropelle ER, Osorio-Costa F, Rossato FA, Vercesi AE, Saad MJ, Carvalheira JB. Metformin amplifies chemotherapy-induced AMPK activation and antitumoral growth. Clin Cancer Res. 2011 Jun 15;17(12):3993-4005. doi: 10.1158/1078-0432.CCR-10-2243. Epub 2011 May 4. PMID 21543517